CLINICAL TRIAL: NCT07023887
Title: EXERT-BCHC: Prospective Study of EXErcise Regimens After Treatment for Breast Cancer for Hypertrophy and Conditioning
Brief Title: Prospective Study of EXErcise Regimens After Treatment for Breast Cancer for Hypertrophy and Conditioning
Acronym: EXERT-BCHC
Status: Recruiting | Type: Observational
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Colin Champ, MD, Principal Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Other Study IDs: 2025-076-SG
Record Dates: First submitted 2025-06-05; First posted 2025-06-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cancer; Breast Cancer
Keywords: exercise
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 6-12-25 Training Regimen — A conditioning regimen involving three exercises performed consecutively with minimal rest. Includes 4-6 repetitions at 4-0-1-0 tempo, 10-12 repetitions at 3-0-1-0 tempo, and 20-25 repetitions at 2-0-1-0 tempo.
Other: 8x8 Training Regimen — A conditioning regimen optimizing high volume with short rest periods. Six exercises are performed consecutively with a 2-0-1-0 tempo and no rest between sets.
Other: 5/5/5 Cluster Set Training Regimen — A hypertrophy regimen where an individual performs 5 repetitions at a tempo of 4 seconds during the eccentric movement of the exercise, while performing the concentric motion in 1 second then resting for 20 seconds and repeating the sequence two additional times to total three clusters of 5 repetitions.
Other: Double Training Regimen — A hypertrophy regimen adding an additional set of lesser repetitions for a specified exercise at the end of a tri-set of exercises.

SUMMARY:
This study investigates the impact of four standard of care, monitored group exercise regimens (resistance training) on conditioning and hypertrophy in women previously treated for breast cancer. The study will compare two conditioning regimens (6-12-25 and 8x8) and two hypertrophy regimens (5/5/5 cluster sets and double training) to assess changes in VO2 max, muscle mass, and fat mass.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-89 years
2. Women prescribed exercise as a Standard of Care
3. Women with a biopsy proven diagnosis of ductal carcinoma in situ (DCIS) or invasive carcinoma of the breast
4. Women must have undergone treatment for breast cancer, including one or more of the following: surgery, radiation therapy, chemotherapy, immunotherapy, or hormonal therapy.
5. Women undergoing active chemotherapy are not allowed on study. Immunotherapy or targeted agent usage is allowed.
6. Women with > 6 months of resistance training experience under expert guidance by a CSCS

Exclusion Criteria:

1. Any current treatment with cytotoxic chemotherapy for breast cancer
2. Inability to safely engage in group sessions of resistance training as deemed by study Pl
3. Severe arthritic, joint, cardiovascular, or musculoskeletal condition deemed by Pl to be unsafe to engage in resistance training
4. Beta blocker or GLP-1 inhibitor medications
5. Pregnant women
6. Males

Ages: 20 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited via convenience sampling from the Study Investigators' practice patient population, referrals from other physicians' practices, or identifiable medical record review (e.g., EPIC).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in VO2 max | Measured monthly during the 5-month exercise program at weeks 4, 8, 12, 16, and 20.
  Change in maximal oxygen consumption (VO2 max) measured during and after each exercise regimen.
Change in Muscle and Fat Mass | Baseline, at the completion of the 5-month exercise program (Week 20), and monthly during the exercise program at weeks 4, 8, 12, and 16.
  Change in muscle mass and fat mass in pounds as measured by InBody 970.
Change in Muscle and Fat Mass | Baseline, at the completion of the 5-month exercise program (Week 20), and monthly during the exercise program at weeks 4, 8, 12, and 16.
  Change in muscle mass and fat mass in pounds as measured by ultrasound.

SECONDARY OUTCOMES:
Change in Hand Grip Strength | Baseline, at the completion of the 5-month exercise program (Week 20), and monthly during the exercise program at weeks 4, 8, 12, and 16.
  Measurement of hand grip strength using a dynamometer to assess upper body strength and function.
Change in Psychology Questionnaire Scores | Baseline, at the completion of the 5-month exercise program (Week 20), and monthly during the exercise program at weeks 4, 8, 12, and 16.
  Assessment of psychological well-being, including confidence, motivation (intrinsic & extrinsic), anxiety, and depression, using a Psychological Screen for Strength Training questionnaire. The responses to the variables will be calculated. The rating scale will be calculated 0-3. Not at all (0), some of the time (1), most of the time (2), and all the time (3).

CONTACTS AND LOCATIONS:
Overall Officials: Colin Champ, Principal Investigator — AHN Radiation Oncology
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request the investigators plan to share unidentified data